CLINICAL TRIAL: NCT01373203
Title: The Role of Fibrocytes in Acute Lung Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Kuan-Jen Bai, Division of Pulmonary & Critical Care Medicine
Other Study IDs: 99077
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Acute Lung Injury(ALI)
Keywords: Acute Lung Injury(ALI)
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The important character of acute lung injury (ALI) is alveolar capillary membrane damage caused by different diseases, such as sepsis, trauma and shock. One of the important pathological stages is the varying degrees of interstitial fibrosis and semi-permeable alveolar membrane fibrosis. It has been proved that CXCL12/SDF-1 (stromal cell-derived factor-1) induces fibrocyte migration, and promotes fibrosis progression. Study indicated that inhibition of TLR4 receptor signaling pathway improves fibrosis progression induced by ALI, however, the role of fibrocyte in ALI is still unclear. The fibrocytes was significantly increased in asthmatic patients with pulmonary fibrosis, which companies with increased CTGF expression. Therefore, this project assumes that fibrocyte will differentiation to fibroblast/myofibroblast in patient with acute lung injury, which in turn leads to progression of fibrosis. The central hypothesis of this project is that peripheral progenitor cell fibrocytes play an important role in alveolitis caused by acute lung injury. The overall objective of this project is to study the role of fibrocytes in acute lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Acute Lung Injury patients
* Above 20 years old
* Bilateral lung infiltrates
* PaO2/FiO2<300mmHg
* PCWP<18mmHg

Exclusion Criteria:

* Pregnant women
* Under 20 years old
* Hb<8.0mg/dl

Min Age: 20 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Lung Injury patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Jen Bai, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan